CLINICAL TRIAL: NCT06230588
Title: A Phase I Clinical Trial to Evaluate the Safety, Tolerability, and Pharmacokinetic Characteristics of TQH3906 Capsules in Healthy Volunteers
Brief Title: A Clinical Trial of TQH3906 Capsules in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TQH3906-I-01
Record Dates: First submitted 2024-01-21; First posted 2024-01-30 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-04

CONDITIONS: Psoriasis
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQH3906 capsule (Experimental): TQH3906 capsule for oral administration as a single or multiple dose for 7days.
  Interventions: Drug: TQH3906 capsule
- TQH3906 placebo capsule (Placebo Comparator): TQH3906 placebo capsule for oral administration as single dose or multiple dose for 7days.
  Interventions: Drug: TQH3906 placebo

INTERVENTIONS:
Drug: TQH3906 capsule — TQH3906 is a kinase inhibitor.
  Arms: TQH3906 capsule
Drug: TQH3906 placebo — Placebo Comparator
  Arms: TQH3906 placebo capsule

SUMMARY:
This study was divided into three parts: single and multiple dosing and food effect study, which were designed to evaluate the safety and tolerability of TQH3906 capsules administered in single or multiple dose escalation in healthy adult subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects aged 18-55 years (including 18 and 55 years), regardless of gender.
* Males weighing ≥ 50 kg, females weighing ≥ 45 kg, with a body mass index (BMI) of 19-26 kg/m2 (included).
* Be in good health with no abnormalities of clinical significance according to medical history, clinical symptoms, vital signs, physical examination, 12-lead electrocardiogram, chest radiographs, abdominal ultrasound, and laboratory tests
* Have a full understanding of the study, participate in the trial voluntarily, and have signed a written informed consent form.
* Subjects (including partners) are willing to voluntarily use appropriate and effective contraception from screening until 3 months after the last dose of study drug.

Exclusion Criteria:

* Pregnant, lactating women.
* Previous history or current cardiac, endocrine, metabolic, renal, hepatic, gastrointestinal, dermatologic, infectious, hematologic, neurologic, or psychiatric disorders/abnormalities, or related chronic illnesses, or acute illnesses, which the investigator assesses as contraindicated for participation in the trial.
* Have a QTc > 450 ms in males and > 470 ms in females at screening, or whose Electrocardiograph (ECG) is unsuitable for Concentration QT (C-QT) measurement (at the discretion of the investigator).
* The presence of risk factors and history of tip-twist ventricular tachycardia including, but not limited to: unexplained syncope, long QT syndrome, heart failure, or clinically significant abnormal laboratory tests (including hypokalemia, hypercalcemia, or hypomagnesemia) identified at Screening.
* Presence of abnormal serum virology at screening;

  1. Active hepatitis, or hepatitis B surface antigen (HBsAg) positive, or Hepatitis C virus (HCV) antibody positive;
  2. Positive for Human immunodeficiency virus (HIV) antibody at the screening stage, or previous history of HIV infection;
  3. Positive antibodies to Treponema pallidum in screening.
* Presence of active tuberculosis during the Screening Period, or being a close household contact of a patient with untreated active tuberculosis, or having a positive tuberculosis interferon gamma release assay (TB-IGRA) by laboratory examination.
* A history of severe bacterial, fungal or viral infection requiring hospitalization for intravenous antibiotic or antiviral medication within 2 months prior to randomization.
* Live vaccination within 4 weeks prior to randomization or planning to receive a live vaccine during the study.
* The presence of clinically significant infections during the Screening Period, including but not limited to upper respiratory tract infections, lower respiratory tract infections, herpes simplex, herpes zoster, and requiring treatment with antibiotics or antiviral medications.
* A history of severe herpes zoster or herpes simplex infection including, but not limited to, herpes encephalitis, disseminated herpes simplex, and herpes zoster pandemic.
* Use of any systemic cytotoxic or systemic immunosuppressive drug within 6 months prior to randomization, or use of any topical cytotoxic or topical immunosuppressive drug within 4 weeks or 5 half-lives (whichever is longer) prior to randomization.
* Receipt of a biologic or other clinical trial drug within 3 months or 5 half-lives, whichever is longer, prior to randomization.
* Has undergone surgery within 4 weeks prior to randomization or is scheduled to undergo surgery during the study.
* Who has lost or donated more than 400 mL of blood within 4 weeks prior to randomization.
* Who have taken any prescription, over-the-counter, and herbal medications, except vitamin products, within 4 weeks prior to randomization.
* Persons with potential blood collection difficulties and a history of needle and blood sickness.
* Allergy to any of the known components of TQH3906 or any previous history of severe drug allergy.
* History of substance abuse or positive urine drug screen.
* Who have smoked more than 5 cigarettes/day or used an equivalent amount of nicotine or nicotine-containing products in the 3 months prior to randomization, or who are unable to discontinue the use of any tobacco-based products during the trial.
* Those who have chronic alcohol abuse or who have consumed more than 14 units of alcohol per week (1 unit = 360 mL of beer or 45 mL of spirits of 40% alcohol by volume or 150 mL of wine) in the 3 months prior to screening or who are unable to abstain from alcohol for the duration of the trial, or who have a positive breath test for alcohol.
* Have any other valid medical, psychiatric, or social reason that, in the opinion of the investigator, precludes participation in this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2024-02-02 (Actual); Primary Completion 2025-04-27 (Actual); Study Completion 2025-04-27 (Actual)

PRIMARY OUTCOMES:
Adverse events (AE) | Up to 18 days
  Incidence of adverse events (AE)
Serious Adverse Events (SAE) | Up to 18 days
  Incidence of serious adverse events (SAE)
Treatment-emergent adverse events (TEAEs) | Up to 18 days
  Incidence of treatment-emergent adverse events (TEAEs)

SECONDARY OUTCOMES:
Time to peak concentration (Tmax) | Up to 18 days
  The time it takes to reach the peak concentration
Peak concentration (Cmax) | Up to 18 days
  Maximum plasma drug concentration
Area under the blood concentration-time curve | Up to 18 days
  The amount of drug absorbed into the circulation after administration of a single dose can be estimated from the area under the blood concentration-time curve, with Auc in units of concentration * time.
Apparent volume of distribution (Vd/F) | Up to 18 days
  It is the ratio of the amount of drug in the body to the blood concentration of the drug when the drug reaches dynamic equilibrium in the body is called the apparent volume of distribution.
Plasma clearance (CL/F) | Up to 18 days
  It is the sum of drug clearance by the liver and kidneys, etc., i.e., how many volumes of plasma are cleared of drug per unit of time in L/h, or L/(kg-h) if calculated on the basis of body weight.
Plasma elimination half-life (t1/2) | Up to 18 days
  The time required for the concentration of a drug in the blood or the amount of drug in the body to be reduced to 1/2. The time required for absorption, distribution and elimination of half the amount of drug (or blood concentration) in the body becomes the absorption half-life, distribution half-life and elimination half-life, respectively.
Steady-state peaking time (Tmax, ss) | Up to 18 days
  The time required to reach a steady-state peak concentration after administration.
Steady state peak concentration (Cmax, ss) | Up to 18 days
  The steady-state blood drug concentration is a serrated plasma drug concentration curve, with the highest steady-state blood drug concentration being the peak steady-state blood drug concentration.
Steady state valley concentration (Cmin, ss) | Up to 18 days
  The steady-state blood drug concentration is a serrated plasma drug concentration curve, with the lowest steady-state blood drug concentration being the trough of the steady-state blood drug concentration.
Average steady-state blood drug concentration (Cav, ss) | Up to 18 days
  The average concentration reached when the drug concentration reaches a steady state after a continuous given dose of medication.
Area under steady-state blood drug concentration time curve (AUC0- τ) | Up to 18 days
  After a single dose administration, the amount of medication absorbed into the human bloodstream can be estimated using the area under the blood drug concentration time curve, with the unit of Auc being concentration * time.
Accumulation ratio (Rac) | Up to 18 days
  The ratio of the required dose for a single administration to the total dose required for a split administration.
Renal clearance rate (CLr/F) | Up to 18 days
  The ability of both kidneys to completely remove a substance equivalent to several milliliters of plasma within one minute.
INF-γ release | Up to 18 days
  Inhibition efficiency of INF-γ release by TQH3906 in IL-12/IL-18-stimulated peripheral blood mononuclear cells from subjects.
QTcF interval | Up to 18 days
  Effect of TQH3906 on the QTcF interval in healthy subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China